CLINICAL TRIAL: NCT03300895
Title: Effect of Low-volume High-intensity Interval Training on Cardiorespiratory Fitness and Total Body Fat in Overweight Women
Brief Title: High-intensity Interval Training on Cardiorespiratory Fitness in Overweight Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Victor Hugo Arboleda Serna, PhD, MSc, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIIT2-AFIS-UdeA
Record Dates: First submitted 2017-09-28; First posted 2017-10-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (Experimental)
  Interventions: Other: High-intensity interval training
- Moderate-intensity continuous exercise (Active Comparator)
  Interventions: Other: Comparator: Moderate-intensity continuous exercise

INTERVENTIONS:
Other: High-intensity interval training — 21.5 minutes of high-intensity interval exercise at an intensity between 90-95 of HRmax (15x30 s), with recoveries at 50-60% of HRmax (14x60 s). 24 sessions, 3x weekly of walking and running outdoors on a sports field in a supervised manner.
  Arms: High-intensity interval training
Other: Comparator: Moderate-intensity continuous exercise — 30 minutes of continuous exercise at an intensity between 65-75% of HRmax. 24 sessions, 3x weekly of walking and jogging outdoors on a sports field in a supervised manner
  Arms: Moderate-intensity continuous exercise

SUMMARY:
High-intensity interval training (HIIT) is currently considered one of the most effective strategies to improved cardiorespiratory fitness, which is recognized as a protective factor for cardiovascular diseases and metabolic diseases such as overweight and obesity. However, current evidence is still limited and requires clarity (frequency, time per session and intensity) regarding to greater increases attributed to HIIT.

The aim of this study is to compare the effect of a low-volume high-intensity interval training versus a moderate-intensity continuous exercise on maximal oxygen consumption in overweight women 18 to 44 years old.

DETAILED DESCRIPTION:
Thirty-six women will be randomly assigned to one of two aerobic exercise on a real-life setting supervised for a physical activity instructor. The interventions will performed three times a week for ten-weeks (on alternate days).

The first two weeks will correspond to the conditioning period (30 minutes between 55-65% of maximum heart rate (HRmax). From week three, 18 participants will perform 30 minutes of continuous exercise at an intensity between 65-75 % of HRmax, and the remaining 18 will complete 21.5 minutes of interval exercise at an intensity between 90-95% of HRmax, with recoveries between 50-55% of HRmax.

All Participants will be evaluated to measure their maximal oxygen consumption, total body fat, waist circumference, body mass index, systolic blood pressure, diastolic blood pressure, prior to start the interventions and at the end of the program (week 11).

ELIGIBILITY:
Inclusion Criteria:

* Overweight (≥ 25 kg/m-2) women 18 to 44 years.
* Healthy volunteers.
* Perform ≤ 600 Met/min/week.

Exclusion Criteria:

* Perform high-intensity interval exercise in the last six month.
* Smoker.
* History of asthma.
* History of diabetes.
* History of hypertension.
* History of cardiovascular disease.
* History of coronary heart disease.
* Arrhythmias.
* Personal history of surgical procedures in the last three months
* Uncontrolled non-communicable diseases
* Under medical treatment with anticoagulants, beta-blockers, calcium antagonists, bronchodilators, and/or steroids.
* Psychological, neuromotor and/or osteo-muscular conditions that may affect participation in an exercise program.
* Psychoactive drug abuse.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change in maximal oxygen consumption | Baseline and after 10 weeks
  Maximal oxygen consumption will be obtained using a graded exercise test on a treadmill (Trackmaster® model TMX 425C) using a portable K4b2 gas analyzer (Cosmed Inc., IL, USA)

SECONDARY OUTCOMES:
Change in total body fat | Baseline and after 10 weeks
  Total body fat will be obtained using an Omron® HBF-510 (Omron Healthcare, Inc. Bannockburn, IL, USA) bioelectrical impedance machine.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arboleda-Serna VH, Patino-Villada FA, Pinzon-Castro DA, Arango-Velez EF. Effects of low-volume, high-intensity interval training on maximal oxygen consumption, body fat percentage and health-related quality of life in women with overweight: A randomized controlled trial. J Exerc Sci Fit. 2022 Apr;20(2):108-112. doi: 10.1016/j.jesf.2022.01.004. Epub 2022 Feb 4. PMID 35228846